CLINICAL TRIAL: NCT06668662
Title: Comparison of Post-operative Pain After Use of Endo-activator and Conventional Irrigation During Endodontic Treatment in Symptomatic Periapical Periodontitis: a Randomized Control Trial
Brief Title: Comparison of Post-operative Pain After Use of Endo-activator and Conventional Irrigation During Endodontic Treatment in Symptomatic Periapical Periodontitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jinnah Sindh Medical University (Other)
Responsible Party: Principal Investigator, Soha Pirzado, Principle Investigator, Jinnah Sindh Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JSMU/IRB/2023/714
Record Dates: First submitted 2024-10-30; First posted 2024-10-31 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Post Operative Pain; Endodontic Treatment; Apical Periodontitis
Keywords: Conventional irrigation; Endoactivator; Post- operative pain; symptomatic periapical periodontitis; Visual Analogue Scale
MeSH Terms: conditions — Pain, Postoperative; Periapical Periodontitis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- endoactivator (Active Comparator): Endoactivator is an irrigation technique which will help to reduce post-operative pain in patients following endodontic treatment.
  Interventions: Device: Endoactivator
- Conventional irrigation (Active Comparator): Conventional irrigation is an irrigation technique which will help to reduce post-operative pain in patients following endodontic treatment.
  Interventions: Device: Conventional irrigation

INTERVENTIONS:
Device: Endoactivator — Endoactivator is an irrigation technique which will help to reduce post-operative pain in patients following endodontic treatment.
  Arms: endoactivator
Device: Conventional irrigation — Conventional irrigation is an irrigation technique which will help to reduce post-operative pain in patients following endodontic treatment.
  Arms: Conventional irrigation

SUMMARY:
Introduction: The adequate removal of microorganisms, infected or necrotic pulp tissues and complete adequate seal of root canal system along with debridement is key to success of endodontic treatment. The objective of this study was to compare frequency of pain after using Endo Activator and conventional irrigation in patients presenting with symptomatic periapical periodontitis following endodontic treatment by means of Visual Analog Scale.

Methods: This study was designed as single blind, randomized control trial. Sixty patients with symptomatic teeth requiring endodontic canal treatment were recruited by probability random sampling into two groups based on irrigation protocols used during endodontic treatment: conventional needle and endo activator irrigation system. The post-operative pain of patients was recorded via a telephone call at 6 hours, 24 hours, and at 7 days on the visual analogue scale (VAS).

DETAILED DESCRIPTION:
Adequate cleaning of root canal system, along with complete eradication of infected, necrotic pulp remnants, persistent microorganisms, and complete sealing of root canal space is key to successful root canal treatment. Activated irrigation is a method that is used to agitate and increase efficacy of irrigant flow to irregularities of root canal spaces as lateral canals and isthmus by chemo-mechanical or various other energy forms and it is one of the irrigation methods used in this study. It has been shown that EndoActivatorTM system produces the effectual irrigation in all spaces of root canal including as lateral canals, isthmuses and the chances of extrusion of irrigant is less than that compared by means of conventional irrigation methods.Thirty seconds use of activated irrigation solution appeared to be more effective in disinfecting root canal compared with an standard irrigation regimen. The most relevant preferred method of activating the irrigant is by using a non-cutting oscillating ultrasonic tip.

NaOCl is the widely used irrigation solution during chemo-mechanical instrumentation as it has a broad range of antibacterial effect and a high capacity of organic tissue dissolution. It has the dissolution capacity when used in concentrations as low as 2.5%, resulting in decreased antibiofilm effect and removal of organic part of smear layer. Similarly, use of EDTA during the preparation removes the organic part of smear layer resulting in exposure of dentinal tubule and for better penetration of NaOCl for disinfection.1 The same protocol and irrigation techniques were followed in our study to maximize the benefit of NaOCl and EDTA during endodontic treatment.

Many studies have examined effects of different various irrigation methods in relation with endodontic procedures on post-operative pain that corroborate with results of this current study. In this study, working length was determined by use of apex locator i.e. electronic measurement device for root canal length which was then confirmed by digital radiograph. This protocol was followed to ensure that preparation was confined within root canal space, and prevent chances of over instru¬mentation that is considered to be one of those major leading cause of post-operative pain.

The Endoactivator System results in minimal extrusion of irritants and irrigate simulated lateral canals at 4.5 and 2 mm from desired working length as compare to that with conventional methods resulting in better irrigation and decreased post-operative pain among different variables.The highest values of post-operative pain were recorded after 6 hours of treatment that potentially decreased in the follow-up periods until almost disappeared after the time interval of one week. In studies evaluation regarding duration of post-operative pain after root canal treatment was noted in regard with above mentioned aggrement.

Studies by Gondim et al and Topçuoğlu et al also reported lower values of pain in Endovac group com¬pared to conventional needle irrigation showing sig¬nificantly marked results after 6 hours followed by 48 hours-time interval. The chances of extrusion of debris apically was greater resulting in increased level of pain with conventional needle-syringe irrigation due to positive pressure of conventional irrigation.

Nivedhitha S 4 in their study concluded that postoperative pain in patients when irrigation was done by means of endoactivator significantly reduced from 6 hours (35.7 ±17.2) to 7 days (4.8±7.4). Topçuoğlu, concluded that after 24 hours, pain in the conventional irrigation group was higher 3.96± 1.95 while endo activator caused mild pain 2.36±1.32.9 Gündoğar in his study concluded that postoperative pain at 48 hours in conventional irrigation group was 0.23±0.63 while that in the endoactivator group was 0.07±0.37.2 Similarly, in the present study canals irrigated by means of endoactivator reported less post-operative pain as compared to canals irrigated with conventional irrigation.

In the present study, the pain score at 6 hours was 4.82±2.690, while at 24 hours was 3.13±2.62 and reduced significantly at 7 days to 1.55±1.789.

The study is aimed to evaluate comparison related to post-operative pain after use of Endoactivator and conventional irrigation during endodontic treatment in symptomatic periapical periodontitis. The VAS scale is a common acceptable method for measuring postoperative pain in research related to dentistry. This scale was described in detail to the patient before recording their pain intensity on the VAS scale so as to reduce significant chances of errors that patients could make while describing their pain intensity. Therefore, patients were made familiar to the VAS and were assisted accordingly in recording their preoperative and postoperative pain conditions. 20 A recent systematic review by Romualdo et al21 stated that apical extrusion of irrigant was considerably less when using apical negative pressure compared in case of using positive pressure techniques. The conclusive findings elaborated that the negative apical pressure decreases the chances of apical extrusion. In the present study, less pain scores were seen in group of endoactivator as compared to those in conventional irrigation group in first 6 hours. These results may be related to fact that chances of extrusion are less in endoactivator group in comparison to the conventional irrigation group. Tang et al 22 in his study also compared the level of post-endodontic pain after single-visit root canal treatment after 24 hours and after one week time interval. However, level of pain was markedly lower in ultrasonic groups compared to the conventional irrigation group at 24 hours and one week after the procedure.

In the first 6 hours after treatment, the greatest post-operative pain scores were seen in both groups, while subsequent observation time points at 24 hours and 7 days showed significant reduction in pain level in both the study groups. Studies that have evaluated postoperative pain after endodontic treatment have reported similar results. 1,4 Pak and White4 in a systematical review concluded that the prevalence of pain diminished from 40% at 24 hours post-endodontic treatment to 11% at the 7th post-operative day.

One of the strengths of this study was random allocation of patients to groups to minimize confounders. Single operator carrying out all the procedures helped to avoid technical errors and standardize the endodontic procedure. Standard protocols for root canal treatment were adhered to in both the study groups for effective root canal treatment to ensure that the post-operative pain could be attributed only to the difference in irrigation protocols.

Despite of certain strengths, the present study focused primarily on vital pulp of single-rooted teeth with fully formed apices, treated in single visit. Therefore, these results may not directly apply to cases involving multi-rooted teeth or immature apices. Moreover, pain is often difficult to measure and can be attributed to multiple variables, so the pinning only one specific cause of pain is quite difficult. In future, studies can be carried out on multirooted teeth with necrotic pulp, treated in multiple visits to evaluate the effect of endoactivator irrigation or other sonic irrigation methods to assess their effect on post endodontic pain incidence.

CONCLUSION:

This study found that intensity and severity of post-operative pain occurring in patients presenting with symptomatic periapical periodontitis was significantly reduced by use of endoactivator when used with 2.5% NaOCl 7 days after single-visit endodontic treatment.

ELIGIBILITY:
Inclusion Criteria: complaints of pain in the maxillary or mandibular single rooted teeth requiring root canal treatment.

* Patients not taking any sedative or analgesics medication 48 hours prior to presenting to the dental clinic
* The teeth that were included were tender to percussion and palpation but had a sound periodontium and no inflammatory exudate or pus drainage.

Exclusion Criteria:

* Patients with any systemic diseases,
* retreatment cases,
* or teeth with calcified canals were excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Comparison of post-operative pain after use of Endo-activator and conventional irrigation during endodontic treatment in symptomatic periapical periodontitis: a randomized control trial. | 6 hours, 24 hours, and at 7 days
  Introduction: The adequate removal of microorganisms, infected or necrotic pulp tissues and complete adequate seal of root canal system along with debridement is key to success of endodontic treatment. The objective of this study was to compare frequency of pain after using Endo Activator and conventional irrigation in patients presenting with symptomatic periapical periodontitis following endodontic treatment by means of Visual Analog Scale.
  Methods: This study was designed as single blind, randomized control trial .Sixty patients with symptomatic teeth requiring endodontic canal treatment were recruited by probability random sampling into two groups based on irrigation protocols used during endodontic treatment: conventional needle and endo activator irrigation system. The post-operative pain of patients was recorded via a telephone call at 6 hours, 24 hours, and at 7 days on the visual analogue scale (VAS).
Endoactivator | The patients were contacted via telephone after 6 hours, 24 hours and 7 days to ask and record their postoperative pain on visual analogue scale that consist of 10cm line anchored by 1 denoting mild and 10 being most severe.
  conventional endodontic needle 4 mL of 2.5% NaOCl was delivered into pulp chamber and then an Endoactivator tip (size #15.02) (DENTSPLY/ Tulsa Dental Specialties, OK) was placed loosely 2 mm short of working length, and activated at 20000 Hz in each canal, moving in a constant in and out motion. The NaOCl was agitated for one minute with approximately 2-3 mm vertical strokes.
Conventional irrigation | The patients were contacted via telephone after 6 hours, 24 hours and 7 days to ask and record their postoperative pain on visual analogue scale that consist of 10cm line anchored by 1 denoting mild and 10 being most severe.
  by placing the needle 2 mm short of desired working length, 4 mL of 2.5% NaOCl was placed into each canal for 40 secs with an approximate flow rate of 0.1 mL/s.

CONTACTS AND LOCATIONS:
Locations (1):
- Sindh Institute of Oral Health Sciences Jinnah Sindh Medical University Karachi, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] 1. Salim A, Darrag A, Ghoneim W. Post-Operative Pain after Single-Visit Endodontic treatment using different root canal irrigation activating techniques. Egypt Dent J. 2021;67(4):3719-30.